CLINICAL TRIAL: NCT02226172
Title: A Phase 2, Double-blind, Randomized Safety And Efficacy Study Of Glasdegib (Pf-04449913) Versus Placebo In Patients With Myelofibrosis Previously Treated With Ruxolitinib
Brief Title: Single-Agent Glasdegib In Patients With Myelofibrosis Previously Treated With Ruxolitinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1371013; SMOI (Other: Alias Study Number); 2014-000933-21 (EudraCT Number); 2014-001048-40 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2018-12

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Primary myelofibrosis; Secondary myelofibrosis; PMF; PET-MF; PPV-MF; Ruxolitinib resistant or intolerant; previously treated myelofibrosis; smoothened inhibitor; oral; single agent.
MeSH Terms: conditions — Primary Myelofibrosis | interventions — glasdegib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Oral daily dose of glasdegib (PF-04449913) 100 mg tablet in a continuous regimen of 28-day cycles.
  Interventions: Drug: Glasdegib (PF-04449913)
- Arm B (Placebo Comparator): Oral daily dose of placebo 100 mg tablet in a continuous regimen of 28-day cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glasdegib (PF-04449913) — Oral daily dose of glasdegib (PF-04449913) 100 mg tablet in a continuous regimen of 28-day cycles.
  Arms: Arm A
Drug: Placebo — Oral daily dose of placebo 100 mg tablet in a continuous regimen of 28-day cycles.
  Arms: Arm B

SUMMARY:
A lead-in cohort of ~20 patients with primary or secondary myelofibrosis previously treated with 1 or more Janus kinase inhibitors enrolled to single-agent glasdegib to evaluate safety and tolerability. Following the lead-in, a phase 2, double blind, 2-arm study, randomized 2:1 to oral single-agent glasdegib versus placebo in 201 patients resistant or intolerant to ruxolitinib.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of primary MF (PMF) or secondary MF (PET-MF and PPV-MF) as per WHO 2008 criteria.
* Lead-in cohort: resistant or intolerant to 1 or more Janus kinase inhibitors (licensed or experimental).
* Randomized cohort: resistant or intolerant to prior ruxolitinib therapy. Documentation by the Investigator that the patient has exhausted available treatment options (eg, resistant or intolerant to hydroxyurea, etc).
* Spleen 5 cm below the inferior left costal margin as measured by manual palpation.
* Active symptomatic MF as defined by the screening MPN-SAD patient-reported instrument requiring a severity score of at least 5 on one symptom, or a severity score of ≥ 3 on at least two of the symptoms (on a 0 to 10 scale).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2, or 3.
* Adequate organ function, demonstrated by the following laboratory values:

  1. Absolute Neutrophil Count 75 x 10(9)/L;
  2. Platelet count >50 x 10(9)/L with no evidence of bleeding and not requiring platelet transfusions;
  3. Serum creatinine <1.5 x upper limit of normal (ULN) or estimated creatinine clearance 60 mL/min (as calculated using the standard method of the institution);
  4. Serum amylase or lipase <1.5 x ULN;
  5. Aspartate aminotransferase and alanine aminotransferase values 3.0 x ULN (or 5x ULN in the case of patients with MF accompanied by hepatic extramedullary hematopoiesis, as manifested by any degree of hepatomegaly).
  6. Total bilirubin values <1.5 x ULN unless the bilirubin is principally unconjugated (in the context of hemolysis) or there is documented Gilbert's disease.
  7. Serum electrolyte values < Grade 2 (sodium, potassium, calcium, phosphorous and magnesium), per CTCAE v.4.03.
* Recovery to Grade 1 from all clinically significant adverse events related to prior MF therapy, including transplant-related toxicities.
* More than 2 months out from allogenic hematopoietic stem cell transplant prior to randomization.
* Must be able to undergo MRI of abdomen (spleen and liver). Patients who are contra indicated for MRI may be enrolled and evaluated by CT scan at the discretion of the Sponsor.
* 18 years of age.
* Male subjects able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use two highly effective methods of contraception throughout the study and for 90 days after the last dose of assigned treatment.

Exclusion criteria:

* Prior treatment with a licensed or experimental smoothened inhibitor.
* Randomized cohort only: Prior treatment with a Janus kinase inhibitor other than ruxolitinib.
* Other anti-cancer therapy up to 14 days prior to enrollment, with the exception of hydroxyurea, which can be given up to 4 days prior to enrollment.
* Splenic irradiation 3 months prior to enrollment.
* History of congenital long QT syndrome, or a baseline >470 msec QTcF abnormality (average of the triplicate reading).
* Evidence of significant cardiac disease, for example: symptomatic cardiac heart failure (CHF, NYHA class 3), complete bundle branch block, significant atrial or ventricular tachyarrhythmias and any unstable cardiac arrhythmias requiring medication.
* History of myocardial infarction or unstable angina within 6 months prior to enrollment.
* Uncontrolled inflammatory bowel disease, peptic ulcer disease or history of significant gastro intestinal bleeding within 6 months of enrollment.
* Any condition requiring chronic use of moderate/high dose steroids (equivalent to 10 mg QD prednisone).
* Hematopoietic growth factor receptor agonists (eg, erythropoietin (Epo), granulocyte colony stimulating factor, romiplostim, eltrombopag within 28 days of enrollment.
* Currently active malignancy (other than MF). Prior malignancies are allowed so long as there is no evidence of disease recurrence within the last 2 years (with the exception of fully excised, non-complicated basal cell carcinoma which can have been active within the prior 2 years, and certain localized, non-invasive fully excised skin, cervical, breast, prostate or bladder tumors).
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH]).
* Active, uncontrolled bacterial, fungal or viral infection, including hepatitis B, hepatitis C, known human immunodeficiency virus or acquired immunodeficiency syndrome related illness.
* Active graft versus host disease (GVHD) with other than grade 1 skin involvement or GVHD requiring immunosuppressive treatment.
* Uncontrolled disseminated intravascular coagulation.
* Current (including their administration within 3 days prior to study entry) use or anticipated need for food or drugs that are strong CYP3A4 inhibitors.
* Current use or anticipated requirement for drugs that are known strong CYP3A4/5 inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (15):
  - Mayo Clinic Building - Phoenix, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UCSD Medical Center Clinical Laboratory - La Jolla, La Jolla, California
  - University of California San Diego (UCSD) Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center- Hillcrest, San Diego, California
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Herbert Irving Comprehensive Cancer Center-Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Huntsman Cancer Institute-University of Utah, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Japan (4):
  - Kobe University Hospital, Kobe, Hyōgo
  - Osaka University Hopsital, Suita-Shi, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371013&StudyName=PF-04449913%20Single-Agent%20In%20Patients%20With%20Myelofibrosis%20Previously%20Treated%20With%20a%20Janus%20Kinase%20Inhibitor

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 2 cohorts were involved lead-in and randomized cohort. Lead-in cohort was followed by randomized cohort. Though the drug was considered safe and tolerable in Myelofibrosis, but a key secondary efficacy outcome measure was not met. Therefore, continuation into the randomized cohort did not proceed.
Groups:
- Glasdegib Lead-in: Glasdegib administered orally at a daily starting dose of 100 mg on a continuous regimen of 28-day cycles.
Period: Overall Study
Arm/Group | Glasdegib Lead-in
Started | 21
Completed | 4
Not Completed | 17
Not completed — Participant refused further follow-up | 4
Not completed — Other | 5
Not completed — Death | 1
Not completed — Study terminated by sponsor | 1
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Spleen Volume Reduction (SVR) ≥35% as Measured by Magnetic Resonance Imaging (MRI)/Computed Tomography (CT) Scan at Week 24 in the Randomized Cohort
Description: The double blind, randomized, placebo controlled phase of the study was not enrolled after the study was terminated early so no data were collected to assess this endpoint.
Time Frame: Week 24
Population: FAS included all participants in the randomized Phase 2 component of the study who were randomized with study drug assignment designated according to initial randomization.
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Treatment -Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Lead-in Cohort
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose of study drug (up to Week 131) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants
  AEs | 21
  SAEs | 5

3. Primary Outcome: Number of Participants With Treatment Emergent Treatment -Related Adverse Events (AEs) and Serious Adverse Events (SAEs): Lead-in Cohort
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose of study drug (up to Week 131) that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator. AEs included both serious and non-serious adverse event.
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants
  AEs | 19
  SAEs | 5

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03: Lead-in Cohort
Description: AE was untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE was AE resulting in any outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability; congenital anomaly.Treatment-emergent were events between first dose of study drug and up to 28 days after last dose of study drug (up to Week 131) that were absent before treatment or that worsened relative to pretreatment state.AE were assessed according to maximum severity grading based on NCI CTCAE Version 4.03.Grade 1=mild; Grade 2=moderate; within normal limits. Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening or disabling; urgent intervention indicated; Grade 5=death. Only categories with at least 1 participant with event were reported.
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants
  Grade 3 or 4 | 14
  Grade 5 | 1

5. Primary Outcome: Number of Participants With Laboratory Abnormalities: Lead-in Cohort
Description: Abnormality: hematology: hemoglobin less than (<)0.8*lower limit of normal(LLN), platelets <0.5*LLN greater than (>)1.75*upper limit of normal(ULN), white blood cell count(WBC) <0.6* LLN >1.5* ULN,lymphocytes, total neutrophils<0.8* LLN >1.2* ULN, band Cells, basophils, eosinophils, monocytes >1.2*ULN, blast cells >1.0*ULN. Coagulation: activated partial thromboplastin time, prothrombin international ratio >1.1* ULN. Liver function: bilirubin >1.5*ULN, AST, ALT,lactate dehydrogenase,alkaline phosphatase >3.0*ULN, protein,albumin <0.8* LLN >1.2* ULN. Renal:blood urea nitrogen,creatinine >1.3*ULN,uric acid >1.2*ULN.Electrolytes: sodium <0.95*LLN >1.05*ULN, potassium, chloride, calcium, magnesium <0.9* LLN >1.1*ULN,phosphate <0.8* LLN >1.2* ULN.Chemistry: glucose <0.6*LLN >1.5*ULN,creatine kinase >2.0*ULN, amylase,lipase >1.5*ULN.Urinalysis: protein, blood >1.0*ULN,red blood cells,WBC >=20,epithelial cells >=6,casts,granular casts,hyaline >1,cellular casts,crystals>=1,bacteria >20.
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants | 21

6. Primary Outcome: Number of Participants With Laboratory Test Abnormalities According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 Grade 3 and Above Hematological Test Abnormalities: Lead-in Cohort
Description: Anemia (grade [g]1:< LLN to 10 gram per deciliter [g/dL],g2:<10 to 8g/dL,g3:<8g/dL, g4:lifethreatening); platelet (g1:<LLN to 75*10^3/millimeter[mm]^3, g2:<75*10^3/mm^3 to 50*10^3/mm^3, g3:<50*10^3/mm^3 to 25*10^3/mm^3, g4:<25*10^3/mm^3); lymphopenia (g1:<LLN to 8*10^2/mm^3, g2:<8*10^2 to 5*10^2/mm^3, g3:<5*10^2 to 2*10^2/mm^3, g4:<2*10^2/mm^3);neutrophil (Absolute) (g1:<LLN to 15*10^2/mm^3, g2:<15*10^2 to 10*10^2/mm^3, g3:<10*10^2 to 5*10^2/mm^3, g4:<5*10^2/mm^3); white blood cell count(g1:<LLN to 3*10^3/mm^3, g2:<3*10^3 to 2*10^3/mm^3, g3:<2*10^3 to 1*10^3/mm^3, g4:<1*10^3/mm^3); hemoglobin (g1:increase in hemoglobin level >0 to 2 g/dL above ULN or above baseline if baseline is above ULN, g2:increase in hemoglobin level>2 to 4g/dL above ULN or above baseline if baseline is above ULN,g3: increase in hemoglobin level>4 g/dL above ULN or above baseline if baseline is above ULN).
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants
  Grade 3 | 3
  Grade 4 | 2

7. Secondary Outcome: Percentage of Participants Achieving SVR ≥35% as Measured by Magnetic Resonance Imaging/Computed Tomography Scan at Week 24 in the Lead-in Cohort
Description: MRI (CT scan may have been permitted if MRI was contraindicated) of the spleen and the liver was performed at baseline, then every 12 weeks while the participant was on treatment. The same method of assessment used at baseline was used for the duration of the trial to ensure consistency. Spleen volume was assessed by a central, independent blinded reader.
Time Frame: Week 24
Population: Lead-in Analysis Set - included all participants treated in the lead-in portion of the study. Only participants who remained on treatment at Week 24 underwent MRI/CT scan.
Measure: Number; unit: Percentage of participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 6
Percentage of participants | 0

8. Secondary Outcome: Percentage of Participants Achieving ≥50% Reduction From Baseline in Total Symptom Score (TSS) as Measured by the Myeloproliferative Neoplasm-Symptom Assessment Diary (MPN-SAD) at Week 24 in the Lead-in Cohort
Description: The MPN-SAD assessed the impact of 9 myelofibrosis symptoms, at their worst, over the past 7 days and over the past 24 hours on a scale of 0 (absent) to 10 (worst imaginable). The 9 symptoms are early satiety, abdominal discomfort, inactivity, night sweats, pruritus, bone pain, pain below the ribs on the left-hand side, fatigue and shortness of breath. The TSS is the sum of the individual scores, excluding inactivity and shortness of breath. The TSS at Week 24 is the average of the daily total scores from the last 28 days of symptom scores immediately prior to Week 24. A higher score indicates worse symptoms.
Time Frame: Week 24
Population: Lead-in Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Percentage of participants | 4.8 [1.2 to 30.4]

9. Secondary Outcome: Monthly Mean Change From Baseline in Overall Total Symptom Score (TSS) in the Lead-in Cohort
Description: as for outcome 8
Time Frame: Weeks 12, 24, 36 and 48
Population: Lead-in Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Score on a scale
  Monthly mean change at Week 12: number analyzed (Participants) | 13
  Monthly mean change at Week 12 | -2.74 (14.07)
  Monthly mean change at Week 24: number analyzed (Participants) | 6
  Monthly mean change at Week 24 | -4.95 (5.78)
  Monthly mean change at Week 36: number analyzed (Participants) | 1
  Monthly mean change at Week 36 | -4.11 (NA) — No standard deviation was calculable since n=1.
  Monthly mean change at Week 48: number analyzed (Participants) | 2
  Monthly mean change at Week 48 | -8.39 (11.52)

10. Secondary Outcome: Percentage of Participants Achieving Anemia Response (Transfusion Dependent Versus Independent) in the Lead-in Cohort
Description: Anemia response was defined as transfusion-independent participants with a ≥20 gram per liter (g/L) increase in hemoglobin (Hb) level where baseline Hb level was <100 g/L, or baseline transfusion-dependent patients becoming transfusion-independent post-baseline. Transfusion dependency before the start of study treatment was defined as transfusions of ≥6 units of packed red blood cells in the 12 weeks prior to start of study treatment, for a final pre-treatment Hb of <85 g/L. In addition, the most recent transfusion episode must have occurred in the 28 days prior to study enrollment. Response in transfusion-dependent patients required absence of any packed red blood cell transfusions during any consecutive rolling 12-week interval during the treatment phase, capped by a Hb level of ≥85 g/L.
Time Frame: Baseline to end of treatment
Population: Lead-in Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Percentage of participants
  Transfusion independent ≥20 g/L Hb increase: number analyzed (Participants) | 17
  Transfusion independent ≥20 g/L Hb increase | 5.9
  Transfusion dependent: number analyzed (Participants) | 4
  Transfusion dependent | 0

11. Secondary Outcome: Maximum Observed Glasdegib Plasma Concentration (Cmax), Minimum Glasdegib Plasma Concentration Observed Prior to the Next Dose (Cmin), and Average Observed Glasdegib Plasma Concentration (Cavg) in the Lead-in Cohort
Description: Cmax was the highest plasma concentration of glasdegib observed directly from the plasma concentration data. Cmin was the lowest plasma concentration of glasdegib observed directly from the plasma concentration data. Cavg was the average concentration at steady state estimated using non-compartmental pharmacokinetic (PK) analysis.
Time Frame: Cycle 1, Day 15
Population: PK Parameter Analysis Population - included all enrolled participants treated who had at least 1 of the PK parameters of interest and were dose compliant (at steady state for glasdegib ).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 19
nanograms per milliliter (ng/mL)
  Cmax | 996.8 (45)
  Cmin | 191.9 (68)
  Cav: number analyzed (Participants) | 17
  Cav | 548.0 (50)

12. Secondary Outcome: Area Under the Glasdegib Plasma Concentration Versus Time Profile at the End of a Dosing Interval (AUCtau) in the Lead-in Cohort
Description: AUCtau was the area under the glasdegib plasma concentration-time profile from time zero to the end of the dosing interval (24 hours) estimated by non-compartmental PK analysis using the linear/log trapezoidal method.
Time Frame: Cycle 1, Day 15
Population: PK Parameter Analysis Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 17
ng·hr/mL | 13150 (50)

13. Secondary Outcome: Time to Reach Cmax (Tmax) in the Lead-in Cohort
Description: Tmax was the time of the first occurrence of Cmax observed directly from the plasma concentration data.
Time Frame: Cycle 1, Day 15
Population: PK Parameter Analysis Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 19
Hours | 1.02 [0.483 to 4.00]

14. Secondary Outcome: Percentage of Participants Achieving SVR ≥50% as Measured by MRI/CT Scan at Week 24 in the Randomized Cohort
Description: as for outcome 1
Time Frame: Week 24
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

15. Secondary Outcome: Monthly Mean Change From Baseline in Overall TSS in the Randomized Cohort
Description: as for outcome 1
Time Frame: Weeks 12, 24, 36 and 48
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants Achieving Anemia Response (Transfusion Dependent Versus Independent) in the Randomized Cohort
Description: as for outcome 1
Time Frame: Baseline to end of treatment
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

17. Secondary Outcome: Participant Reported Outcomes of Health Related Quality of Life and Health Status in the Randomised Cohort
Description: as for outcome 1
Time Frame: Baseline to end of treatment
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

18. Secondary Outcome: Median Duration of SVR in the Randomized Cohort
Description: as for outcome 1
Time Frame: Baseline to end of treatment
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

19. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival in the Randomized Cohort
Description: as for outcome 1
Time Frame: Baseline to end of treatment
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

20. Secondary Outcome: Glasdegib PK Parameters in the Randomized Cohort
Description: as for outcome 1
Time Frame: Cycle 1, Day 15
Population: PK Parameter Analysis Population
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

21. Secondary Outcome: Psychometric Validation of the MPN-SAD in the Randomised Cohort
Description: as for outcome 1
Time Frame: Baseline to end of treatment
Population: FAS
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

22. Secondary Outcome: Number of Participants With Treatment -Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Randomized Cohort
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state.
Time Frame: Baseline up to Week 131
Population: The double blind, randomized, placebo controlled phase of the study was not enrolled as the study was terminated early so, no data were collected to assess this outcome measure.
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Participants With Treatment Emergent Treatment -Related Adverse Events (AEs) and Serious Adverse Events (SAEs): Randomized Cohort
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to Week 131
Population: as for outcome 22
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

24. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) According to Maximum Severity: Randomized Cohort
Description: AE was untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE was AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AE were assessed according to maximum severity grading based on NCI CTCAE Version 4.03.Grade 1=mild; Grade 2=moderate; within normal limits. Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening or disabling; urgent intervention indicated; Grade 5=death.
Time Frame: Baseline up to Week 131
Population: as for outcome 22
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

25. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Randomized Cohort
Description: Abnormality: hematology: hemoglobin less than (<)0.8*lower limit of normal(LLN), platelets <0.5*LLN >1.75*upper limit of normal(ULN), white blood cell count(WBC) <0.6* LLN greater than (>)1.5* ULN,lymphocytes, total neutrophils<0.8* LLN >1.2* ULN, band Cells, basophils, eosinophils, monocytes >1.2*ULN, blast cells >1.0*ULN. Coagulation: activated partial thromboplastin time, prothrombin international ratio >1.1* ULN. Liver function: bilirubin >1.5*ULN, AST, ALT,lactate dehydrogenase,alkaline phosphatase >3.0*ULN, protein,albumin <0.8* LLN >1.2* ULN. Renal:blood urea nitrogen,creatinine >1.3* ULN,uric acid >1.2* ULN.Electrolytes: sodium <0.95*LLN >1.05*ULN, potassium, chloride, calcium, magnesium <0.9* LLN >1.1*ULN,phosphate <0.8* LLN >1.2* ULN.Chemistry: glucose <0.6*LLN >1.5*ULN,creatine kinase >2.0*ULN, amylase,lipase >1.5*ULN.Urinalysis: protein, blood >1.0*ULN,red blood cells,WBC >=20,epithelial cells >=6,casts,granular casts,hyaline >1,cellular casts,crystals>=1,bacteria >20.
Time Frame: Baseline up to Week 131
Population: as for outcome 22
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

26. Primary Outcome: Number of Participants With Laboratory Test Abnormalities According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 Grade 3 and Above Chemistry Test Abnormalities: Lead-in Cohort
Description: ALT/AST g1:>ULN 3*ULN, g2:>3-5*ULN, g3:>5 20*ULN, g4:>20*ULN); Alkaline Phosphatase (g1:>ULN 2.5*ULN,g2:>2.5-5*ULN, g3:>5 20*ULN, g4:>20*ULN); Creatinine (g1:>ULN-1.5*ULN,g2:>1.5-3*ULN, g3:>3 6*ULN, g4:>6*ULN);hyperglycemia (g1:>ULN-160,g2:>160 250, g3:>250 500, g4:>500mg/dL);bilirubin(total) (g1:>ULN-1.5*ULN, g2:>1.5-3*ULN, g3:>3 10*ULN,g4:>10*ULN);hypoglycaemia (g1:<LLN-55,g2:<55-40, g3:<40 30,g4:<30mg/dL); hyperkalemia (g1:>ULN-5.5,g2:>5.5-6, g3:>6 7,g4:>7mmol/L);hypokalemia (g1:<LLN-3,g2:<LLN-3, g3:<3 2.5, g4:<2.5mmol/L);hypermagnesemia (g1:>ULN-3,g3:>3 8, g4:>8mg/dL);hypocalcemia (g1:<LLN-8,g2:<8-7, g3:<7-6, g4:<6mg/dL); hypercalcemia (g1:>ULN-11.5,g2:>11.5-12.5, g3:>12.5-13.5, g4:>13.5mg/dL); hypomagnesemia (g1:<LLN-1.2,g2:<1.2-0.9,g3:<0.9-0.7, g4:<0.7mg/dL); hyponatremia (g1:<LLN-130,g3:<130-120, g4:<120mmol/L);hypoalbuminemia (g1:<LLN-3,g2:<3 2,g3:<2, g4:lifethreatening);hypophosphatemia (g1:<LLN-2.5,g2:<2.5-2, g3:<2-1, g4:<1mg/dL).
Time Frame: Baseline up to Week 131
Population: All participants treated in the lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 21
Participants
  Grade 3 | 5
  Grade 4 | 1

27. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities By Maximum Severity: National Cancer Institute Common Terminology Criteria for Adverse Event (Version 4.0) Grade 3 and Above Hematological Test Abnormalities: Randomized Cohort
Description: Anemia g1:< LLN to 10 g/dL, g2:<10 to 8g/dL, g3:<8g/dL, g4:lifethreatening); platelet (g1:<LLN to 75*10^3/mm^3, g2:<75*10^3/mm^3 to 50*10^3/mm^3, g3:<50*10^3/mm^3 to 25*10^3/mm^3, g4:<25*10^3/mm^3); lymphopenia (g1:<LLN to 8*10^2/mm^3, g2:<8*10^2 to 5*10^2/mm^3, g3:<5*10^2 to 2*10^2/mm^3, g4:<2*10^2/mm^3);neutrophil (absolute) (g1:<LLN to 15*10^2/mm^3, g2:<15*10^2 to 10*10^2/mm^3, g3:<10*10^2 to 5*10^2/mm^3, g4:<5*10^2/mm^3); white blood cell count (g1:<LLN to 3*10^3/mm^3, g2:<3*10^3 to 2*10^3/mm^3, g3: <2*10^3 to 1*10^3/mm^3, g4:<1*10^3/mm^3); hemoglobin(g1:increase in hemoglobin level>0 to 2 g/dL above ULN or above baseline if baseline is above ULN, g2: increase in hemoglobin level>2 to 4g/dL above ULN or above baseline if baseline is above ULN, g3:increase in hemoglobin level>4 g/dL above ULN or above baseline if baseline is above ULN).
Time Frame: Baseline up to Week 131
Population: as for outcome 22
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

28. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities By Maximum Severity: National Cancer Institute Common Terminology Criteria for Adverse Event (Version 4.0) Grade 3 and Above Chemistry Test Abnormalities: Randomized Cohort
Description: ALT/AST g1:>ULN 3*ULN, g2:>3-5*ULN, g3:>5 20*ULN, g4:>20*ULN); Alkaline Phosphatase (g1:>ULN 2.5*ULN, g2:>2.5-5*ULN, g3:>5 20*ULN, g4:>20*ULN);Creatinine (g1:>ULN-1.5*ULN, g2:>1.5-3*ULN, g3:>3 6*ULN, g4:>6*ULN);hyperglycemia (g1:>ULN-160,g2:>160 250, g3:>250 500,g4:>500mg/dL); bilirubin(total) (g1:>ULN-1.5*ULN, g2:>1.5-3*ULN, g3:>3 10*ULN,g4:>10*ULN); hypoglycaemia (g1:<LLN-55, g2:<55-40, g3:<40 30, g4:<30mg/dL); hyperkalemia (g1:>ULN-5.5,g2:>5.5-6, g3:>6 7,g4:>7mmol/L); hypokalemia (g1:<LLN-3,g2:<LLN-3,g3:<3 2.5, g4:<2.5mmol/L); hypermagnesemia (g1:>ULN-3,g3:>3 8,g4:>8mg/dL); hypocalcemia (g1:<LLN-8,g2:<8-7, g3:<7-6, g4:<6mg/dL); hypercalcemia (g1:>ULN-11.5,g2:>11.5-12.5, g3:>12.5-13.5, g4:>13.5mg/dL);hypomagnesemia (g1:<LLN-1.2,g2:<1.2-0.9, g3:<0.9-0.7,g4:<0.7mg/dL); hyponatremia (g1:<LLN-130,g3:<130-120, g4:<120mmol/L);hypoalbuminemia (g1:<LLN-3,g2:<3-2, g3:<2, g4:lifethreatening);hypophosphatemia (g1:<LLN-2.5,g2:<2.5-2,g3:<2-1,g4:<1mg/dL).
Time Frame: Baseline up to Week 131
Population: as for outcome 22
Arm/Group | Glasdegib Lead-in
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 131
Description: An event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event. All participants treated in the lead-in portion of the study. It was the analysis population for all analyses on the lead-in portion of the study.
Arm/Group | Glasdegib Lead-in
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glasdegib Lead-in (N=21)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Confusional state (Psychiatric disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glasdegib Lead-in (N=21)
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Fatigue (General disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Electrocardiogram QT prolonged (Investigations) | 3
Lipase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 3
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Investigators will, on request, remove any previously undisclosed Confidential Information (other than the Study results themselves) before disclosure.